CLINICAL TRIAL: NCT01993277
Title: A Comparator Trial Evaluating Three Neuromodulation Technologies' Effectiveness in Early Recovery From Substance Abuse Disorders as Compared to Relaxation Therapy
Brief Title: Evaluating Neuromodulation Technologies in Early Recovery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Behavioral Health of the Palm Beaches (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2013-11-16; First posted 2013-11-25 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Depression; Anxiety; Insomnia
MeSH Terms: conditions — Depression; Anxiety Disorders; Sleep Initiation and Maintenance Disorders | interventions — Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Fischer Wallace Stimulator (Active Comparator): 30 20-minute sessions of the Fischer Wallace Stimulator administered twice-per-day within a 3-week time-frame;
  Interventions: Device: Fischer Wallace Stimulator
- Nexalin Brain Stimulator (Active Comparator): 15 40-minute sessions of Nexalin Brain Stimulator adminsitered once-per-day within a 3-week time-frame
  Interventions: Device: Nexalin Brain Stimulator
- DAVID Delight Stimulator (Active Comparator): 15 40-minute sessions of the DAVID Delight administered once-per-day within a 3-week time-frame
  Interventions: Device: David Delight Stimulator
- Relaxation Therapy (Active Comparator): 15 40-minute relaxation therapy sessions once-per-day within a 3-week time-frame
  Interventions: Behavioral: Relaxation Therapy

INTERVENTIONS:
Device: Nexalin Brain Stimulator
  Arms: Nexalin Brain Stimulator
Device: Fischer Wallace Stimulator
  Arms: Fischer Wallace Stimulator
Device: David Delight Stimulator
  Arms: DAVID Delight Stimulator
Behavioral: Relaxation Therapy
  Arms: Relaxation Therapy

SUMMARY:
The study is an open-label comparative effectiveness clinical trial evaluating the impact of three neuromodulation treatment devices to improve the mental health and sobriety status of recovering substance abuse patients. We intend to enroll 200 patients to give us a sufficient number of subjects for the planned comparisons. Following informed consent and baseline assessment, patients will be randomly assigned to receive either 1) 15 40-minute sessions of Nexalin Brain Stimulator, a cranial electrical stimulation (CES) device, once-per-day within a 3-week time-frame; 2) 30 20-minute sessions of the Fischer Wallace Stimulator, another CES device, twice-per-day within a 3-week time-frame; 3) 15 40-minute sessions of the DAVID Delight, an audio-visual stimulation device (AVS), once-per-day within a 3-week time-frame; OR 4) the control-group condition of 15 40-minute relaxation therapy sessions once-per-day within a 3-week time-frame. All subjects will then be reassessed at the end of the 3 weeks of treatment and again 1, 3, and 6 months later. In addition to the assigned treatments, all patients will also receive the standard array of services that are provided by Behavioral Health of the Palm Beaches (BHOPB) including as clinically appropriate, psychiatric medication management and Eye Movement Desensitization Response (EMDR) therapy. Patients diagnosed with Post Traumatic Stress Disorder (PTSD) are assessed to determine their suitability for EMDR and if suitable, will receive 2 or more EMDR sessions. Patients without PTSD do not receive EMDR therapy.

ELIGIBILITY:
Inclusion Criteria:

Adults between the ages of 18 and 75 in early recovery from a substance abuse disorder.

Exclusion Criteria:

The exclusion criteria are patients diagnosed with 1) an uncontrolled seizure disorder, 2) a psychotic disorder with currently active features (e.g., paranoia), 3) a dissociative identity disorder, 4) a manic episode within the past month, 5) patients with a pace-maker or implanted vagal nerve stimulator, patients prescribed Subocone, Subutext, &/or any psychostimulant medication (e.g., Alderol, Concerta, Focalin, Metadate, Vyvance, etc.) since these medications interfere with the ability of these neuromodulation devices' ability to have the intended effect on patients, and 7) pregnant woman.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-06 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
The Quick Inventory of Depressive Symptoms-Self-Report (QIDS-SR) | Change in baseline depressive symtpoms, after 3 weeks of treatment, and 1, 3, and 6 months followup
State-Trait Anxiety Inventory (STAI) | Change in baseline anxiety symtpoms, after 3 weeks of treatment, and 1, 3, and 6 months followup
Pittsburgh Sleep Scale (PSS) | Change in baseline insomnia symtpoms, after 3 weeks of treatment, and 1, 3, and 6 months followup
16-item Quality of Life Enjoyment and Satisfaction Questionnaire (QLES) | Change in baseline quality of life, after 3 weeks of treatment, and 1, 3, and 6 months followup

SECONDARY OUTCOMES:
Brief Substance Craving Scale (BSCS) | Change in baseline craving intensity after the 5th, 10th, and 15th treatment sessions

CONTACTS AND LOCATIONS:
Overall Officials: Tammy Malloy, LCSW, Principal Investigator — Behavioral Health of the Palm Beaches; Jodi Star, M.D., Principal Investigator — Behavioral Health of the Palm Beaches; Kate Reynolds, MSW, Principal Investigator — Behavioral Health of the Palm Beaches
Locations (1):
- Behavioral Health of the Palm Beaches, North Palm Beach, Florida, United States